CLINICAL TRIAL: NCT06329050
Title: The Effects of Losartan on Attention Control: An Eye-tracking Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAM_lab_eyetracking_02
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Eye-tracking; Losartan
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Losartan tablet(50 mg)
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Administration of Losartan tablets(50 mg)
  Other Names: Cozaar
  Arms: Losartan group
Drug: Placebo — Administration of Placebo tablets
  Other Names: Placebo treatment
  Arms: Placebo group

SUMMARY:
The main aim of the present study is to investigate the effects of orally administered Losartan on bottom-up and top-down attentional control to socio-emotional stimuli by combining a validated saccade/antisaccade eye-tracking paradigm with a randomized between-subject placebo-controlled pharmacological trial design.

DETAILED DESCRIPTION:
Animal models and initial findings in humans suggest that the angiotensin II antagonist Losartan may have neuroprotective effects and could potentially enhance cognitive functions, including valence-specific attention and regulatory control. Within this context the present study aims to examine whether angiotensin II blockade via Losartan modulates top-down and bottom-up attentional control towards socio-affective stimuli. To this end, healthy individuals will undergo a double-blind, between-subjects, placebo-controlled pharmaco-eye-tracking experiment and receive a single oral dose of Losartan (50 mg) or placebo before performing a saccade/anti-saccade task 90 minutes after administration. The task paradigm will encompass social (happy, angry, fearful, sad and neutral faces) and non-social (oval) stimuli to examine general as well as social and emotion-specific effects of oral losartan.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects who volunteer to participate and are able to fully understand and agree with this study by written informed consent.

Normal or corrected-normal version

Exclusion Criteria:

* History of neuropsychiatric diseases.
* History of cardiac disease, including arrhythmias, aortic stenosis, or congestive heart failure; history of syncope or unexplained loss of consciousness.
* History of hepatic diseases, including cholestasis, biliary obstructive disease, or severe liver dysfunction.
* History of renal diseases, including renal stones or renal failure.
* History of hyponatremia(Serum sodium <135mmol/L) or hyperkalemia (Serum potassium>5.5mmol/L); history of diabetes mellitus or diabetes insipidus
* Known hypersensitivity or allergic reaction to any medication or hormone; strong allergic reaction to food.
* Infections such as COVID-19 or influenza, or unexplained fever.
* Subjects with hypertension (BP ≥130/80mmHg) or hypotension (BP ≤ 90/60mmHg).
* History of alcohol or drug abuse; smoker (≥ 10 cigarettes or ≥ 3 cigars or ≥ 3 pipes/day); smoker using e-cigarettes.
* Blood donation (≤ 1 month prior to administration).
* Take oral contraceptives or receive hormonal medications in the three months prior to the experiment.
* Pregnant or breastfeeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Saccade/antisaccade latency difference between social and non-social stimuli after losartan administration | 90 minutes - 120 minutes after treatment
  Comparison between social-specific saccade/antisaccade latencies (in milliseconds) between the losartan and placebo treatment conditions.
Error rate of saccade/antisaccade for social versus non-social stimuli after losartan administration | 90 minutes - 120minutes after treatment
  Comparison between social-specific error rates of saccade/antisaccade between the losartan and placebo treatment conditions.

SECONDARY OUTCOMES:
Saccade/antisaccade latency for different facial emotions after losartan administration | 90 minutes - 120 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade latencies (in milliseconds) between the losartan and placebo treatment conditions.
Error rate of saccade/antisaccade for different facial emotions after losartan administration | 90 minutes - 120 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade error rates between the losartan and placebo treatment conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China